CLINICAL TRIAL: NCT00701155
Title: Observational, Safety Study in Subjects Using Insulin Detemir for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus
Brief Title: Observational Study to Evaluate the Safety While Using Levemir®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1953
Record Dates: First submitted 2008-06-13; First posted 2008-06-19 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the actual clinical evaluation
  Other Names: Levemir®

SUMMARY:
This study is conducted in Africa. The aim of this observational study is to evaluate the incidence of serious adverse drug reactions while using insulin Levemir® under normal clinical practice conditions in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* After the physician decision has been made to use insulin detemir, any subject with Type 1 or Type 2 diabetes mellitus is eligible for the study, including newly-diagnosed subjects who have never received insulin or an insulin analogue before. The selection of the subjects will be at the discretion of the individual physician.

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit;
* Subjects currently being treated with insulin detemir;
* Subjects who previously enrolled in this study
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients
* Pregnancy, breast-feeding, the intention to become pregnant or judged not to be using adequate contraceptive measures. (Adequate contraceptive measures are an intrauterine device, oral contraceptives and barrier methods)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 or 2 diabetes patients
Sampling Method: Non-Probability Sample
Enrollment: 3593 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious ADRs incl. major hypoglycemias | after 24 weeks

SECONDARY OUTCOMES:
Number of serious adverse events | after 24 weeks
Number of all adverse events | after 24 weeks
Weight changes | after 24 weeks
HbA1c | after 24 weeks
Subgroup analysis of hypoglycemias | after 24 weeks
Number of all hypoglycemic events | in the 4 weeks preceding the visits at 12 weeks and 24 weeks.
Variability in fasting Blood Sugar and average plasma glucose levels | after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Giza, Egypt

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com